CLINICAL TRIAL: NCT05396040
Title: School Studies Within the EuCARE Horizon Europe Research Project (EUCARE-SCHOOLS Study)
Brief Title: School Studies Within the EuCARE Horizon Europe Research Project (EuCARE-SCHOOLS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Euresist Network GEIE (Other)
Collaborators: University of Salento (Other); Istituto Europeo di Oncologia (Other); University of Milan (Other); University of Lisbon (Other); University of Cologne (Other); Hospital Regional de Alta Especialidad "Dr. Juan Graham Casasus" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EuCARE-SCHOOLS
Record Dates: First submitted 2022-05-18; First posted 2022-05-27 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-08

CONDITIONS: STUDENTS

STUDY DESIGN:
Intervention Model Description: The study will enrol 440 classes (around 8800 students, teachers and other personnel) from 2 countries, randomised to Lolli-Methode or SoC. Samples from pools will be regularly collected and tested using PCR-based techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LOLLI METHODE (Experimental): regular screening with pooled saliva tests (Lolli-Method)
  Interventions: Procedure: LOLLI METHODE
- STANDARD OF CARE (No Intervention): STANDARD OF CARE

INTERVENTIONS:
Procedure: LOLLI METHODE — WEEKLY SCREENING WITH POOLED SALIVA PCR TEST
  Arms: LOLLI METHODE

SUMMARY:
In this clinical trial, the aim is to determine if regular screening with pooled saliva tests (Lolli-Method) is useful to support school opening and to reduce clusters and attack rates in schools, compared with the standard of care (SoC) regular surveillance based on symptoms and contact tracing by public health departments.

DETAILED DESCRIPTION:
In this clinical trial, it will be determined if regular screening with pooled saliva tests (Lolli-Method) is useful to support school opening and to reduce clusters and attack rates in schools, compared with the standard of care (SoC) regular surveillance based on symptoms and contact tracing by public health departments. A multicenter cluster randomised interventional study will be set-up to evaluate the efficacy and applicability of the Lolli-Methode. The study will enrol 440 classes (around 8800 students, teachers and other personnel) from 2 countries, randomised to Lolli-Methode or SoC. Samples from pools will be regularly collected and tested using PCR-based techniques. Test results will be combined with questionnaires filled in by children, parents and schools teachers and principals, concerning social distancing measures implemented and psychological impact of the preventive measures applied during the pandemic. A thorough data analysis will then be performed to understand the applicability of Lolli-Methode to reduce SARS-COV-2 transmission in schools, including incidence, attack rates and cluster analysis. On the other hand, mobility changes and psychological outcomes will be analysed and compared with variables related to SARS-COV-2 transmission. By the end of this study, it will be identified and characterised the applicability of the Lolli-Methode for SARS-COV-2 surveillance, as well as the impact of pandemic preventive measures on children.

An ancillary observational study will be carried out on a different population of schools to study the prevalence of SARS-COV-2, frequencies and size of clusters and attack rates in schools, compared with those of previous waves; to compare the effectiveness of different preventive measures adopted in different schools; to investigate psychological issues in students and teachers related to the pandemic's containment measures.

ELIGIBILITY:
Inclusion Criteria:

* Kindergartens and school-age children from public or private schools .
* Enrolled children may be students of classes that have expressed their consent to participate
* School personnel of participating schools
* Householders of participating children
* Informed consent (for minors the informed consent will be signed by parents or legal guardians) .
* For minors: will to participate.

Exclusion Criteria:

* No informed consent by schools or children, or the adult participant
* Suspicion of acute COVID-19 infection:

In case of unknown respiratory infection, no presence of symptoms for at least 48 hours. In case of confirmed SARS-COV-2 infection: inclusion at the earliest 21 days from PCR-positive diagnosis after the onset of potential symptoms and no presence of symptoms for at least 48 hours (according to Standard of Care).

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3373 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Frequencies of clusters | up to 18 months
  Frequencies of clusters in classrooms in which pooled saliva tests (Lolli-Method) are performed in association with standard contact-tracing protocols, compared with classrooms in which SoC protocols are applied.
Number of participating classes | up to 18 months
  Number of classes and of students in the classes that accept to participate in the Lolli-Methode study, if asked, during time

SECONDARY OUTCOMES:
Transmission/prevalence of SARS-COV-2 in schools by variants | up to 18 months
  Transmission/prevalence of SARS-COV-2 in schools by variants, by assessing the proportion of students/staff with positive SARS-COV-2 test identified by pooled saliva tests (Lolli-Method)
Psychological status of children | up to 18 months
  Psychological status of children during coronavirus pandemics: negative and positive feeling during confinement, worries and expectations about school resumption as evaluated by questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCESCA INCARDONA, Study Chair — EURESISTE NETWORK GEIE
Locations (5):
- Italy (3):
  - DISTEBA, Università del Salento, Lecce, Apulia
  - IEO Istituto Europeo di Oncologia Research Hospital and Treatment Centre, Milan, Lombardy
  - Università statale di Milano, Dipartimento di Scienze Biomediche e Cliniche L. Sacco, Milan, Lombardy
- Hospital Regional de Alta Especialidad Dr. Juan Graham Casasus, Villahermosa, Tabasco, Mexico
- Global Health and Tropical Medicine; Instituto de Higiene e Medicina Tropical, Universidade Nova de Lisboa (UNL), Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
The study is part of a project funded by the European Commission and the project agreement with the Commission affirms that the data and the results will be public
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after the Study end no time limit was fixed
Access Criteria: request to the study coordinator or to he project partners
URL: https://eucareresearch.eu/

REFERENCES:
- [Background] Ozer EA, Simons LM, Adewumi OM, Fowotade AA, Omoruyi EC, Adeniji JA, Dean TJ, Zayas J, Bhimalli PP, Ash MK, Godzik A, Schneider JR, Mamede JI, Taiwo BO, Hultquist JF, Lorenzo-Redondo R. Coincident rapid expansion of two SARS-CoV-2 lineages with enhanced infectivity in Nigeria. medRxiv [Preprint]. 2021 Jul 2:2021.04.09.21255206. doi: 10.1101/2021.04.09.21255206. PMID 33880483
- [Background] Robson F, Khan KS, Le TK, Paris C, Demirbag S, Barfuss P, Rocchi P, Ng WL. Coronavirus RNA Proofreading: Molecular Basis and Therapeutic Targeting. Mol Cell. 2020 Sep 3;79(5):710-727. doi: 10.1016/j.molcel.2020.07.027. Epub 2020 Aug 4. PMID 32853546
- [Background] Sekine T, Perez-Potti A, Rivera-Ballesteros O, Stralin K, Gorin JB, Olsson A, Llewellyn-Lacey S, Kamal H, Bogdanovic G, Muschiol S, Wullimann DJ, Kammann T, Emgard J, Parrot T, Folkesson E; Karolinska COVID-19 Study Group; Rooyackers O, Eriksson LI, Henter JI, Sonnerborg A, Allander T, Albert J, Nielsen M, Klingstrom J, Gredmark-Russ S, Bjorkstrom NK, Sandberg JK, Price DA, Ljunggren HG, Aleman S, Buggert M. Robust T Cell Immunity in Convalescent Individuals with Asymptomatic or Mild COVID-19. Cell. 2020 Oct 1;183(1):158-168.e14. doi: 10.1016/j.cell.2020.08.017. Epub 2020 Aug 14. PMID 32979941
- [Background] Singh J, Samal J, Kumar V, Sharma J, Agrawal U, Ehtesham NZ, Sundar D, Rahman SA, Hira S, Hasnain SE. Structure-Function Analyses of New SARS-CoV-2 Variants B.1.1.7, B.1.351 and B.1.1.28.1: Clinical, Diagnostic, Therapeutic and Public Health Implications. Viruses. 2021 Mar 9;13(3):439. doi: 10.3390/v13030439. PMID 33803400
- [Derived] Raimondi S, Gandini S, Rubio Quintanares GH, Abecasis A, Lopalco PL, D'Ecclesiis O, Chiocca S, Tomezzoli E, Cutica I, Mazzoni D, Amparo N, Pingarilho M, Carmagnola D, Dellavia C, Zuccotti G, Ronchini C, Bellerba F, Dewald F, Kaiser R, Incardona F; Eucare WP4. European Cohorts of patients and schools to Advance Response to Epidemics (EuCARE): a cluster randomised interventional and observational study protocol to investigate the relationship between schools and SARS-CoV-2 infection. BMC Infect Dis. 2023 Jan 3;23(1):1. doi: 10.1186/s12879-022-07947-6. PMID 36597074
- See also: Otte im Kampe et al, Surveillance of COVID-19 school outbreaks, Germany, March to August 2020, Eveline Otte im Kampe et al., Eurosurveillance, Sept 2020 — https://www.eurosurveillance.org/content/10.2807/1560-7917.ES.2020.25.38.2001645